CLINICAL TRIAL: NCT04823468
Title: Effect of Oral Nutritional Supplements From the Beginning of Radiotherapy on Body Weight Loss of Patients With Nasopharyngeal Carcinoma and Its Cost-Utility Analysis: A Prospective Multicenter Randomized Controlled Trial
Brief Title: Effect of Oral Nutritional Supplements on Body Weight Loss of Patients With Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinsheng Hong (Other)
Collaborators: Fujian Cancer Hospital (Other Government); The Second Affiliated Hospital of Fujian Medical University (Other); The Nanping First Affiliated Hospital of Fujian Medical University (Unknown); Quanzhou First Hospital (Other); Fujian Medical University Union Hospital (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Hunan Cancer Hospital (Other); Jiangxi Provincial Cancer Hospital (Other); 900 Hospital of Joint Logistics Support Force of PLA (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor-Investigator, Jinsheng Hong, Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FYYY-FLK-202001
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma; Nutritional Support
Keywords: Nasopharyngeal Carcinoma; Nutritional Support; Chemoradiotherapy; Dietary Supplements; Body Weight; Cost-Effectiveness Analysis
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Body Weight | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In addition to conventional dietary instruction and individualized nutritional counselling, patients were given additional ONS (Abbott®Ensure of 55.8 g tid) from the beginning to the end of radiotherapy.
  Interventions: Dietary Supplement: Abbott®Ensure; Radiation: Intensity Modulated Radiation Therapy; Drug: cisplatin
- Control group (Other): Conventional dietary instruction and individualized nutritional counselling from the beginning to the end of radiotherapy.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: cisplatin

INTERVENTIONS:
Dietary Supplement: Abbott®Ensure — Abbott®Ensure: 55.8 g each time, three times a day, from the beginning to the end of radiotherapy
  Arms: Experimental group
Radiation: Intensity Modulated Radiation Therapy — The prescribed dose was 68-76 Gy to Planning target volume of the primary tumor (PTVnx), 66-70 Gy to Planning target volume of the cervical lymph node (PTVnd), 60-64 Gy to planning target volume 1 (PTV1), and 50-54 Gy to planning target volume 2 (PTV2) in 30-33 fractions. The details of dose limits for organs at risk were based on the study 0225 from The Radiation Therapy Oncology Group (RTOG 0225).
Drug: cisplatin — 80-100 mg/m² cisplatin given intravenously every 3 weeks concurrently with radiotherapy.

SUMMARY:
Concurrent chemoradiotherapy(CCRT) is the principal treatment for nasopharyngeal carcinoma(NPC). Studies have shown that malnutrition is very common in patients with NPC after chemoradiotherapy. Malnutrition can lead to weight loss, treatment interruption, prolonged stay in hospital, increased treatment costs, reduced tolerance to anti-tumor therapy, reduced quality of life and shortened survival time. Nutritional intervention can improve the nutritional status, reduce treatment-related toxicity and improve the survival of patients with NPC.

The first choice of nutritional intervention is oral nutritional supplements(ONS). Some retrospective studies with small samples have found that early nutritional intervention can reduce weight loss and severe oral mucositis in patients with NPC, compared with late nutritional intervention. Therefore, the investigators proposed the hypothesis that ONS from the beginning of radiotherapy can reduce the nutritional impairment, treatment-related toxicity and treatment costs of patients with NPC, and improve their quality of life. The aim of this multicenter randomized controlled clinical trial is to evaluate the efficacy and cost utility of ONS from the beginning to the end of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma;
* All genders, range from 18-70 years old;
* Clinical stage II-IVa according to the 8th edition of the Union for International Cancer Control/American Joint Committee on Cancer (UICC/AJCC) staging system;
* Patient-Generated Subjective Nutrition Assessment (PG-SGA) score ≤8;
* Main organ functions test should be satisfied the following conditions: (1) Absolute neutrophil count (ANC) ≥1.5×10^9/L; (2) Platelet (PLT) ≥80×10^9/L; (3) Hemoglobin (Hb) ≥90 g/L; (4) Bilirubin < 1.5 times the upper limit of normal value (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times the upper limit of normal value; (5) Creatinine < 1.5 times the upper limit of normal value or creatinine clearance rate >60 ml/min.

Exclusion Criteria:

* Patients whose energy intake is less than 60% of the target energy requirement for 3 days or more;
* Have or are suffering from other malignant tumors;
* Refuse concurrent chemoradiotherapy;
* With diabetics, galactosemia, or sever metabolic diseases or endocrine diseases;
* Cannot take oral or enteral nutrition, including intestinal obstruction, severe short bowel syndrome or high output fistula, or with severe digestive system diseases;
* Known allergic reaction to any component of Abbott®Ensure, or severe allergic constitution;
* Pregnant or lactating women;
* With previous or ongoing clinical trials;
* Refuse to sign inform consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of weight loss > 5% | From time of randomization to the date of radiotherapy ends, up to 7 weeks
  The percentage of patients whose body weight decreased more than 5% over baseline, body weight (in kilograms) are measured at baseline and weekly during the course of radiotherapy

SECONDARY OUTCOMES:
PG-SGA Score | From time of randomization to the date of radiotherapy ends, up to 7 weeks
  The scores assessed by Patient-Generated Subjective Nutrition Assessment (PG-SGA) at baseline and weekly during the course of radiotherapy
Incidence of participants with grade ≥3 oral mucositis | During the course of radiotherapy, up to 7 weeks
  Incidence of grade 3-4 oral mucositis assessed by CTCAE v5.0, evaluated weekly during radiotherapy
Days of radiotherapy interruption | During the course of radiotherapy, up to 7 weeks
  The number of days that radiotherapy was interrupted due to treatment-related toxicity
Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 v3.0 (EORTC QLQ-C30 v3.0) | From time of randomization to the date of radiotherapy ends, up to 7 weeks
  The standard scores assessed by the EORTC QLQ-C30 v3.0 at baseline and the end of radiotherapy.
Increment Cost-Utility Ratio (ICUR） | During the course of chemoradiotherapy, up to 7 weeks
  The Increment cost-utility ratio is used to assess the economics of ONS, which is calculated as incremental cost divided by incremental utility.
Score of EQ-5D-5L questionnaire | During the course of chemoradiotherapy, up to 7 weeks
  The standard scores assessed by the EuroQol- 5 dimension-5 level (EQ-5D-5L ) questionnaire. Collect this questionnaire only in the responsible center.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsheng Hong, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (13):
- China (13):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - 900th hospital of the joint logistics team, PLA, Fuzhou, Fujian
  - The Nanping First Affiliated Hospital of Fujian Medical University, Nanping, Fujian
  - Quanzhou First Hospital Affiliated to Fujian Medical University, Quanzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No